CLINICAL TRIAL: NCT01438645
Title: ScopeGuide-assisted Colonoscopy Versus Conventional Colonoscopy for Improved Endoscopic Performance and Enhanced Patient Experience
Brief Title: ScopeGuide-assisted Colonoscopy Versus Conventional Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Teshima (Other)
Responsible Party: Sponsor-Investigator, Christopher Teshima, Assistant Professor, University of Alberta
Organization: University of Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ScopeGuide 01
Record Dates: First submitted 2011-09-14; First posted 2011-09-22 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Colonic Neoplasms; Iron Deficiency Anemia; Diarrhea
Keywords: Colonoscopy; Colon cancer screening
MeSH Terms: conditions — Colonic Neoplasms; Anemia, Iron-Deficiency; Diarrhea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ScopeGuide-assisted colonoscopy (Experimental): These patients will undergo colonoscopy with the assistance of the Olympus ScopeGuide system.
  Interventions: Device: Olympus ScopeGuide
- Conventional colonoscopy (No Intervention): These patients will undergo colonoscopy identical to that in the intervention arm, except with endoscopes lacking the ScopeGuide system.

INTERVENTIONS:
Device: Olympus ScopeGuide — ScopeGuide-assisted colonoscopy using Olympus CF-H180DL variable-stiffness colonoscopes equipped with ScopeGuide capabilities. ScopeGuide will provide the endoscopist with a 3-dimensional image on the monitor depicting the shape of the colonoscope inside the patient's body as it moves through the colon.
  Other Names: Magnetic endoscopy imaging
  Arms: ScopeGuide-assisted colonoscopy

SUMMARY:
Colonoscopy is an established technology that enables doctors to obtain live video from inside patients' large intestines, which is essential for the diagnosis of numerous intestinal illnesses. It consists of a long, flexible tube fitted with a light-source and small video camera that transmits the images onto a display monitor. The doctor inserts the scope into the anus, moves it into the rectum and then guides it slowly through the entire colon. Because of the various twists and turns that are part of normal bowel anatomy, advancing the scope through the entire colon is not always successful and can become challenging when the scope forms loops inside the abdomen. Unfortunately, there is no way for the doctor to see the shape of the scope inside the body other than what is seen from the video at its front end, and so navigating the colon relies on instinct accumulated with experience and the "feel" of the scope as loops begin to form. This is important because not only can this loop formation cause pain, but it can also increase the likelihood of an incomplete test. Incomplete tests matter because a major reason for performing colonoscopy is colon cancer screening and surveillance; detecting early cancers at treatable stages and looking for polyps that may be pre-cancerous growths. When colonoscopy does not advance through the entire colon, parts are left unexamined where cancer may develop. A new technology called "ScopeGuide" has been developed that uses magnetic coils embedded within the scope to create a 3D image of the shape of the entire scope inside the body that is projected onto the monitor for the doctor to see. This will show if loops are forming and will provide information about how to eliminate loops once they have formed. In this research study, the investigators will compare colonoscopy with the assistance of ScopeGuide to colonoscopy performed in the standard fashion, to see if ScopeGuide results in more successful procedures that are easier for the doctor and more comfortable for patients.

DETAILED DESCRIPTION:
Summary of Research Proposal

Background:

Colon and rectal cancer (CRC) is a leading cause of cancer-related morbidity and mortality in Canada. Colonoscopy is the preferred screening modality for CRC and has been shown to decrease the likelihood of developing CRC as well as CRC-related mortality, particularly through the detection and removal of potentially pre-cancerous polyps, with the aim of preventing colon cancer, and for the diagnosis of early stage CRC that is more likely to be treatable and result in long-term survival. However, recent evidence suggests that colonoscopy has not been as universally protective against CRC as had been previously hoped, particularly for proximal cancers located in the right colon. Theories as to why this might be the case include speculation about altered biology of cancers that develop in the proximal colon and technical issues relating to the performance of colonoscopy itself. In particular, one of the problems is incomplete colonoscopy that fails to examine the entire colon to the cecum, which may occur in 10-20% of cases. Furthermore, from a public health standpoint, a considerable proportion of the population remain averse to undergoing colonoscopy, particularly because of fears of procedure discomfort, decreasing the potential impact for overall CRC reduction. Thus, optimizing the technical performance of colonoscopy and improving its acceptance among patients is important for maximizing the possible benefits to society.

One of the most common reasons for incomplete colonoscopy is excessive internal looping of the endoscope. This looping has also been shown to be the major cause of patient discomfort during the procedure. Experts agree that colonoscopy is most successful at reaching the cecum and most comfortable for patients when the endoscope is kept in a straight position by minimizing loop formation and reducing loops once they have formed. Thus, identification and reduction of endoscope loops is critically important for the successful and comfortable completion of colonoscopy. Over the years, several techniques have emerged to overcome loop formation, including withdrawal of the endoscope with torque, abdominal wall pressure and patient position changes, yet these are all done in a "trial and error" fashion. Despite this limitation, these maneuvers form the cornerstones of current colonoscopy technique. Technological innovations such as smaller caliber "pediatric" colonoscopes and "variable stiffness" colonoscopes with adjustable rigidity have been introduced that have had moderate success in diminishing patient discomfort and increasing rates of colonoscopy completion. Yet despite these efforts to improve colonoscopy practice, the reality is that many procedures are still done poorly. An audit of all colonoscopies performed in Winnipeg from 2004 to 2006 demonstrated a dismal completion rate of only 65%. Thus, something more clearly needs to be done. In an effort to help improve colonoscopy from both the technical standpoint of the endoscopist and also the comfort level of patients, Olympus has redesigned a previously developed real-time imaging system that enables visualization of the shape of the entire endoscope while it is inside the patient's body. This technology, called ScopeGuide (Olympus America, Center Valley, PA), consists of electromagnetic coils embedded within the endoscope that are detected by an external receiver dish, generating a 3D representation of the endoscope that is displayed on a monitor. It is anticipated that by visualizing the entire scope as it moves through the body, endoscopists will gain useful visual information about loop formation and scope position that will enable greater technical success while creating a more comfortable patient experience.

Study Objectives:

The purpose of this project is to perform a randomized, non-blinded colonoscopy study to determine if real time visualization of the colonoscope using the new Olympus ScopeGuide system is superior to conventional colonoscopy for the achievement of endoscopic procedural outcomes and for an improved patient experience in terms of reduced discomfort and decreased sedation requirements.

Methods:

Consecutive patients referred for colonoscopy at the University of Alberta Hospital (UAH) will be considered for study enrollment. Eligible patients who meet the inclusion and exclusion criteria and who provide informed consent will be randomized to undergo conventional colonoscopy or colonoscopy with the assistance of the ScopeGuide system. The control group will use Olympus CF-H180AL variable-stiffness, high-definition colonoscopes that do not differ from the usual procedure and the investigational group will use Olympus CF-H180DL variable-stiffness, high-definition colonoscopes equipped with ScopeGuide capabilities. ScopeGuide will provide the endoscopist with a 3-dimensional image on the monitor depicting the shape of the colonoscope inside the patient's body as it moves through the colon.

The colonoscopy will be performed as clinically indicated, either with or without the aid of the ScopeGuide system. All patients will undergo a purgative bowel preparation followed by an overnight fast prior to their colonoscopy according to standard clinical practice at UAH. At the start of the colonoscopy, all patients will initially be given standardized doses of conscious sedation medications consisting of midazolam 2 mg IV and fentanyl 25 mcg IV. However, the procedure may be initiated without any sedation upon patient request. Additional doses of sedative medications may be given at patient request or when the nurse or physician believes that the patient is uncomfortable. In all cases, the endoscopist will attempt to minimize the formation of loops within the colon and will straighten those loops whenever possible. This will be achieved by conventional methods that rely on "feel" and "instinct" in the control group and will be directed by the ScopeGuide visualization in the investigational group. The endoscopist may use any technical maneuvers deemed necessary to facilitate completion of the procedure, including the application of external abdominal pressure by the nurse, the repositioning of the patient, or tightening of the variable-stiffness setting of the colonoscope. Upon intubation of the cecum, the insertion distance of the colonoscope from the anus to the cecal pole will be recorded as a marker of the straightness of the endoscope. Any abnormalities detected during colonoscope insertion will be more closely inspected, photographed and biopsied during subsequent colonoscope withdrawal. Furthermore, polyps will also be preferentially removed during colonoscope withdrawal, which is the existing standard-of-care. Any diagnostic or therapeutic applications that are required during the colonoscopy are permitted as clinically indicated.

Relevant demographic and clinical information will be recorded prior to the procedure. Additional data regarding procedural metrics, technical maneuvers, and sedation doses will be recorded during the colonoscopy. At the conclusion of the colonoscopy, the endoscopist will rate the procedural difficulty as "usual" or "difficult" and will also note the procedural diagnosis.

After the procedure, the patient will be kept in the post-endoscopy recovery area in the usual fashion. Prior to discharge home from the recovery area, participants will complete a visual analogue scale reflecting their degree of discomfort experienced during the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient 18 years or older.
2. Able to read & write English.
3. Undergoing colonoscopy at University of Alberta Hospital for any indication.

Exclusion Criteria:

1. Colonoscopy performed without prior purgative bowel prep.
2. Patient with active, ongoing lower GI bleeding.
3. Colonoscopy performed to attempt colonic decompression in acute colonic pseudo-obstruction (Ogilvie's syndrome).
4. Colonoscopy for which propofol sedation is required.
5. Inpatient colonoscopy performed by a trainee under staff supervision.
6. Patient with previous colonic surgery.
7. Patient with pacemaker or implantable cardioverter-defibrillator (ICD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sedation Score | 1 day (immediate outcome assessment at time of endoscopy procedure)
  The main efficacy parameter is the amount of sedation used during colonoscopy, expressed as the mean for each group. Since our conscious sedation consists of two different drugs, the doses of each will be converted into a numerical score, such that typical 1 mg dose increments of midazolam and 25 mcg increments of fentanyl will each be assigned a score of '1,' and the two will be added together to give the sedation score.

SECONDARY OUTCOMES:
Patient comfort | 1 day (immediate outcome assessment after recovery from endoscopy procedure)
  Patients wil complete a 10 cm visual analogue pain scale (VAS) that will be converted to a numerical score (0-100) with each number representing 1 mm on the 10 cm VAS from 0 at its left extreme (representing 'no pain') to 100 on its right extreme (representing 'unbearably severe pain'). The mean pain score will then be determined for each of the groups.
Time-to-cecum | 1 day (immediate outcome assessment at time of endoscopy procedure)
  Time from initial insertion of colonoscope until successful intubation of the cecum (min)
Cecal intubation rate | 1 day (immediate outcome assessment at time of endoscopy procedure)
  Proportion of colonoscopy procedures resulting in successful intubation of the cecum.
Ancillary maneuvers to facilitate procedure | 1 day (immediate outcome assessment at time of endoscopy procedure)
  Number of added maneuvers, including abdominal pressure, repositioning of patient, endoscope loop reduction techniques, used to facilitate advancement of endoscope during procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W Teshima, MD FRCPC, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Shah SG, Brooker JC, Williams CB, Thapar C, Saunders BP. Effect of magnetic endoscope imaging on colonoscopy performance: a randomised controlled trial. Lancet. 2000 Nov 18;356(9243):1718-22. doi: 10.1016/S0140-6736(00)03205-0. PMID 11095259
- [Background] Shah SG, Brooker JC, Thapar C, Suzuki N, Williams CB, Saunders BP. Effect of magnetic endoscope imaging on patient tolerance and sedation requirements during colonoscopy: a randomized controlled trial. Gastrointest Endosc. 2002 Jun;55(7):832-7. doi: 10.1067/mge.2002.124097. PMID 12024136
- [Derived] Teshima CW, Zepeda-Gomez S, AlShankiti SH, Sandha GS. Magnetic imaging-assisted colonoscopy vs conventional colonoscopy: a randomized controlled trial. World J Gastroenterol. 2014 Sep 28;20(36):13178-84. doi: 10.3748/wjg.v20.i36.13178. PMID 25278714